CLINICAL TRIAL: NCT04916665
Title: Bridging Intestinal Failure With Teduglutide - a Case Report
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Felix Harpain, Principle Investigator, M.D., Medical University of Vienna
Other Study IDs: 8745632
Record Dates: First submitted 2021-05-30; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome | interventions — teduglutide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Teduglutide — bridging intestinal failure with teduglutide until reconstruction

SUMMARY:
In this case report the investigators present a novel strategy for using teduglutide as a bridging therapy to intestinal reconstruction.

ELIGIBILITY:
Inclusion Criteria:

short bowel syndrome

Exclusion Criteria:

* <18 years

Sex: Male
Age Groups: Child, Adult, Older Adult
Study Population: case report
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
enteral autonomy (complete discontinuation of parenteral support) | 6 months
  observe if enteral autonomy may be achieved before reconstruction

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No